CLINICAL TRIAL: NCT01045356
Title: Pharmacokinetics of Tranexamic Acid (TXA) in Children Undergoing Repair of Congenital Heart Defects Utilizing Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark C. Wesley, MD, Boston Children's Hospital
Other Study IDs: x10-01-0006
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2011-06

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- children less than 2 months old
- children 2 months to 12 months old
- Children > 2 months old and less than or equal to 20 kg

SUMMARY:
The purpose of this study is to measure blood levels of TXA in children having cardiac surgery which requires cardiopulmonary bypass. TXA is used to reduce bleeding during surgery. This study will help determine if the current dosing of TXA results in therapeutic blood levels.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart disease requiring surgical repair with cardiopulmonary bypass

Exclusion Criteria:

* children weighing over 20 kg
* family does not want to participate in the study

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with congenital heart defects having cardiac surgery requiring cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine TXA blood levels in children having cardiac surgery with cardiopulmonary bypass. The current dosing recommendations will be utilized. | multiple times thoughout surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dowd NP, Karski JM, Cheng DC, Carroll JA, Lin Y, James RL, Butterworth J. Pharmacokinetics of tranexamic acid during cardiopulmonary bypass. Anesthesiology. 2002 Aug;97(2):390-9. doi: 10.1097/00000542-200208000-00016. PMID 12151929